CLINICAL TRIAL: NCT03334266
Title: Preventing Early Childhood Obesity, Part 2: Family Spirit Nurture, Prenatal - 18 Months
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 7871
Record Dates: First submitted 2017-10-03; First posted 2017-11-07 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Obesity; Infant Obesity; Mother-Child Relations; Dietary Habits; Breast Feeding; Physical Activity; Childhood Obesity; Feeding Behavior
Keywords: sugar; sweetened; beverages; responsive
MeSH Terms: conditions — Obesity; Pediatric Obesity; Feeding Behavior; Breast Feeding; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Spirit Nurture (FSN) (Experimental): The intervention group (n=169) will receive the Family Spirit Nurture (FSN) + Optimized Standard Care (OSC). The FSN home-visiting module consists of 36, 60-minute lessons delivered by trained local Family Health Coaches (FHCs), from 28 weeks gestation to 18 months postpartum. Lessons focus on three key content domains: 1) promotion of optimal breastfeeding, complementary and responsive feeding across early childhood; 2) promotion of healthy infant/toddler diet and physical activity, as well as reduced screen time and sedentary lifestyle; and 3) promotion of maternal psychosocial well-being, optimization of healthy food/beverage availability and identification/creation of safe play spaces in the home environment.
  Interventions: Behavioral: Family Spirit Nurture (FSN); Other: Optimized Standard Care (OSC)
- Control Program (Other): The control group will receive Injury Prevention Education (IPE) + Optimized Standard Care (OSC). The IPE home-visiting module consists of 8 30-minute lessons delivered by trained local Family Health Liaisons (FHL), from 28 weeks gestation to 18 months postpartum. The lessons will be delivered at the following assessment time points: 36 weeks gestation, 2 weeks, 2 months, 4 months, 6 months, 9 months, 12 months, and 18 months postpartum. Injury prevention lessons focus on injury prevention topics relevant to the participating communities but that will not overlap in anyway with FSN content, including: motor vehicle safety for mothers and children; preventing scald burns; fire safety; child-proofing a home; preventing falls; preventing poisonings; and preventing animal bites.
  Interventions: Other: Injury Prevention Education (IPE); Other: Optimized Standard Care (OSC)

INTERVENTIONS:
Behavioral: Family Spirit Nurture (FSN) — The FSN home-visiting module consists of 36 60-minute lessons delivered by trained local FHCs, from 28 weeks gestation to 18 months postpartum. The lessons focus on three key content domains: 1) promotion of optimal breastfeeding, complementary and responsive feeding across early childhood; 2) promotion of healthy infant/toddler diet and physical activity, as well as reduced screen time and sedentary lifestyle; and 3) promotion of maternal psychosocial well-being, optimization of healthy food/beverage availability and identification/creation of safe play spaces in the home environment.
  Arms: Family Spirit Nurture (FSN)
Other: Injury Prevention Education (IPE) — The control group will receive Injury Prevention Education (IPE). The IPE home-visiting module consists of 8 30-minute lessons delivered by trained local Family Health Liaisons (FHL), from 28 weeks gestation to 18 months postpartum. Injury prevention lessons focus on injury prevention topics relevant to the participating communities, including: motor vehicle safety for mothers and children; preventing scald burns; fire safety; child-proofing a home; preventing falls; preventing poisonings; and preventing animal bites.
  Arms: Control Program
Other: Optimized Standard Care (OSC) — OSC will be available to both in the FSN intervention and control groups. OSC consists of transportation assistance to prenatal and well-baby clinic visits as recommended by the Indian Health Service (IHS) and American Academy of Pediatrics (AAP) and rescue services through linkages to community agencies as needed.

SUMMARY:
This study aims to assess the impact of a home-visiting program, called "Family Spirit Nurture" (FSN), on reducing early childhood obesity in American Indian (AI) children. The FSN intervention targets parent feeding practices, young children's diet and physical activity (PA) and early childhood (0-2 years of age) weight status, all associated with risk for early childhood obesity and, consequently, risk for obesity over the life course. The investigators will also explore whether maternal psychosocial factors (stress, depression and substance use), household food/water security and/or constrained physical activity environments moderate FSN intervention impacts on: mother's feeding behaviors for infants and toddlers; and, children's diets, PA patterns, and weight status. Finally, the investigators will examine how maternal/infant characteristics, diet and behaviors impact the underlying biologic mechanisms of early childhood obesity and whether social and behavioral interventions can impact infant metabolic health. The investigators evaluation will employ a randomized controlled design, in which both the intervention and comparison condition receive assisted transportation to prenatal and well-baby visits (called "Optimized Standard Care"), and the comparison condition also receives potentially beneficial injury prevention education at 8 assessment visits.

Primary Aims:

Efficacy of Family Spirit Nurture (FSN) + Optimized Standard Care (OSC) versus Injury Prevention Education (IPE) + OSC will be assessed for each of the following from birth to 24 months postpartum:

Aim 1. Mothers' implementation of recommended feeding behaviors. Hypothesis 1. FSN + OSC mothers will be more likely to meet breastfeeding and complementary feeding recommendations and engage in responsive parenting/feeding behaviors compared to IPE + OSC mothers.

Aim 2. Children's consumption of healthy diet and physical activity engagement. Hypothesis 2. FSN + OSC children will consume more fruits and vegetables and fewer calories from sugar sweetened beverages (SSB), snacks and desserts, and they will have higher physical activity and reduced screen time/other sedentary activities compared to IPE + OSC children.

Aim 3. Children's weight status. Hypothesis 3. Mean BMI z-scores for FSN + OSC children will be closer to zero (the mean age- and sex- specific BMI z-score for the World Health Organization standard reference population) compared to IPE + OSC children.

DETAILED DESCRIPTION:
Secondary Aims:

Secondary Aim 1. To explore whether maternal psychosocial factors (stress, depression and substance use), and household food/beverage security and/or constrained physical activity environments moderate FSN intervention impacts on: infant and young children's feeding behaviors; and, infant/young children's diets, PA patterns, and weight status.

Secondary Aim 2. To explore how maternal/infant characteristics, diet and behaviors impact the underlying biologic mechanisms of early childhood obesity, and whether social and behavioral interventions can impact infant metabolic health.

Aim 2a. At delivery, examine how measures of infant metabolic health (fasting glucose, insulin, leptin, adiponectin, lipids, and c-reactive protein) are a) correlated with maternal biologic measures of metabolic health (fasting glucose, insulin, leptin, adiponectin, lipids, and c-reactive protein) and b) are impacted by sociodemographic, biological and psychosocial characteristics of mothers at baseline (e.g. age, parity, water/food security, BMI, gestational weight gain, gestational diabetes, depression, perceived stress). Hypothesis: Infant biologic measures of metabolic health will be highly correlated with maternal levels of metabolic health at birth and will vary by maternal baseline characteristics.

Aim 2b. Between delivery and 12 months postpartum, examine how biologic measures of infant metabolic health change in relation to a) maternal biologic measures of metabolic health, b) sociodemographic, biological and psychosocial characteristics of mothers at baseline, and c) maternal/infant behaviors (e.g. responsive feeding practices, infant diet, introduction of sugar-sweetened beverages, early physical activity, etc.). Hypothesis: Biologic measures of infant metabolic health over the first 12 months of life will begin to diverge from maternal levels; and, infant metabolic health between delivery and 12 months postpartum will vary by maternal baseline characteristics and maternal/infant behaviors across study groups.

Aim 2c. Infant metabolic health. Hypothesis: FSN + OSC infants will have better metabolic health (defined by fasting glucose, insulin, leptin, adiponectin, lipid and c-reactive protein levels) at 12 months postpartum compared with IPE + OSC infants.

Secondary Aim 3. To explore how specific community- and tribal level policy, systems, and environmental (PSE) factors affect child feeding practices, healthy weight status, SSB and water consumption, and safe water access on the Navajo Nation.

Aim 3a. Assess the impact of actual and perceived water insecurity on child feeding practices and children's weight and metabolic status. Hypothesis: Participants who do not have or do not trust their household water sources breastfeed less, and feed more SSBs and less water to children, impacting weight and metabolic status at 24 months of life.

Aim 3b. Explore community readiness and political will to address water insecurity among policy, systems, and environmental leaders on the Navajo Nation. Hypothesis: Examination of community- and tribal-level policy, systems, and environmental facilitators and barriers to safe water access will provide key knowledge to promote children's water vs. SSB intake and healthy weight status.

Aim 3c. Compare actual vs. perceived household water safety and determine the distance it takes water insecure households to access safe drinking water. Hypothesis: The distance participants travel to access safe water affects what beverages they feed young children.

Secondary Aim 4. To explore how the COVID-19 pandemic impacted infant/child feeding practices, food and water security, and study participation. Hypothesis: Examination of how the COVID-19 pandemic impacted study outcomes will provide important knowledge about how future home-visiting interventions can best adapt to community-level crises.

The investigators will conduct a randomized 1:1 controlled trial with 338 mothers (ages 14 to 24) and their children (ages 0-24 months) living in the three study sites (2 Navajo; 1 Apache). Assessments in both groups will occur at baseline (< 32 weeks gestation), 36 weeks gestation, delivery (blood sample collection only), 2 weeks, 2 months, 4 months, 6 months, 9 months, 12 months, 18 months, and 24 months postpartum.

Intervention: The intervention group (n=169) will receive the FSN + OSC. OSC consists of transportation assistance to prenatal and well-baby clinic visits as recommended by the Indian Health Service (IHS) and American Academy of Pediatrics (AAP) and rescue services through linkages to community agencies as needed. The FSN home-visiting module consists of 36 60-minute lessons delivered by trained local FHCs, from 28 weeks gestation to 18 months postpartum. The lessons will be delivered bi-weekly from 28 weeks gestation to birth, weekly from birth to 3 months postpartum, bi-weekly from 3 to 6 months postpartum and monthly from 6 to 18 months postpartum. The lessons focus on three key content domains: 1) promotion of optimal breastfeeding, complementary and responsive feeding across early childhood; 2) promotion of healthy infant/toddler diet and physical activity, as well as reduced screen time and sedentary lifestyle; and 3) promotion of maternal psychosocial well-being, optimization of healthy food/beverage availability and identification/creation of safe play spaces in the home environment.

Comparison Condition: The comparison group will receive IPE + OSC. The IPE home-visiting module consists of 8 30-minute lessons delivered by trained local Family Health Liaisons (FHL), from 28 weeks gestation to 18 months postpartum. The lessons will be delivered at the following assessment time points: 36 weeks gestation, 2 weeks, 2 months, 4 months, 6 months, 9 months, 12 months, and 18 months postpartum. Injury prevention lessons focus on injury prevention topics relevant to the participating communities but that will not overlap in anyway with FSN content, including: motor vehicle safety for mothers and children; preventing scald burns; fire safety; child-proofing a home; preventing falls; preventing poisonings; and preventing animal bites.

OSC transportation visits for both the intervention and comparison groups include transportation for up to 6 prenatal visits from 28 weeks gestation to birth and 8 well-baby visits during the first 18 months of life. OSC was selected because it optimizes the standard of care for young mothers and their children within reservation communities, addresses transportation and access barriers, provides beneficial and ecologically-valid services in the participants' settings, and was previously approved and endorsed by Community Advisory Boards and tribal Institutional Review Boards. By providing OSC to both intervention and control groups, the quality and dose of OSC is controlled so differences between study arms can be validly attributed to the FSN intervention. Two hours is allotted for each OSC visit (for transportation and waiting at clinic visit) x 14 visits = 28 hours of obstetric/pediatric care support. OSC visits will also be used to administer maternal self-reports at relevant time points for both study arms.

Both the intervention and comparison condition participants will receive a follow-up assessment at 24 months, but no education sessions will take place with either study group between 18 and 24 months postpartum.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to participate
2. 14 to 24 years old at the time of conception
3. < 32 weeks gestation at the time of enrollment
4. Reside within 1 hour (50 miles) of local Indian Health Service medical facility
5. Willingness to undergo random assignment and participate in all aspects of the study

Exclusion Criteria:

1. Inability to participate in full intervention or evaluation (e.g., planned move, residential treatment, etc.)

Ages: 14 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 259 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Group differences in percentage of mothers who meet breastfeeding and complementary feeding recommendations and percentage of mothers who introduce sugar sweetened beverages over time as assessed by the Child Feeding Assessment. | 2 weeks - 24 months postpartum
  Mothers will be asked questions from an adapted version of the Pre-School-Aged Beverage Intake Questionnaire (BEVQ-15) in addition to items developed by the study team and based on previous studies conducted by the co-investigators. The assessment will be used to assess feeding practices, duration of exclusive and non-exclusive breastfeeding, timing of introduction of complementary foods and types of first foods, and introduction of SSBs among infants/toddlers, including questions about the frequency and amount of child's beverage intake
Group differences in mean scores for infant feeding style subscales assessed using the Infant Feeding Behavior Questionnaire. | 2 months-12 months postpartum
  The Infant Feeding Behavior Questionnaire (IFBQ) (administered at 2, 6, and 12 months postpartum) asks mothers to indicate how often they engage in specific feeding behaviors to assess maternal feeding styles. There are 5 subscales that are used to assess maternal feeding style; Responsive, Forceful, Restrictive, Indulgent, and Uninvolved. There is no total scale score. The assessment is valid and reliable. This 24-item scale is scored with a 3-point Likert scale. A mean score is calculated for each subscale, with a range of 0 to 2. The range of the 3-point Likert scale is as follows: 0 (never), 1 (sometimes), 2 (always). Higher scores reflect higher levels of feeding style indicated by a given subscale. So, for example, for responsive feeding a higher score would be better, and for forceful feeding a higher score would be worse.
Group differences in in mean scores for toddler feeding style subscales assessed using the Toddler Feeding Behavior Questionnaire (TFBQ). | 24 months postpartum
  The TFBQ (administered at 24 months postpartum) asks mothers to indicate how often they engage in specific feeding behaviors to assess maternal feeding styles. There are 5 subscales that are used to assess maternal feeding style; Responsive, Forceful, Restrictive, Indulgent, and Uninvolved. There is no total scale score. The assessment is valid and reliable. This 27-item scale is scored with a 3-point Likert scale. A mean score is calculated for each subscale, with a range of 0 to 2. The range of the 3-point Likert scale is as follows: 0 (never), 1 (sometimes), 2 (always). Higher scores reflect higher levels of feeding style indicated by a given subscale. So, for example, for responsive feeding a higher score would be better, and for forceful feeding a higher score would be worse.
Group differences in children's fruit and vegetable intake, sugar sweetened beverage (SSB) consumption, snacks, and desserts over time. | 6 and 24 months postpartum
  Mothers will be asked questions about child's fruit and vegetable consumption beginning at 6 months postpartum and at all subsequent time points. These items have been added to the standardized 18-item U.S. Department of Agriculture (USDA) food security survey. Fruit and vegetable (F&V) consumption will be measured by asking mothers how much and how often her child eats F&Vs and whether she feels she is able to provide her child with the F&Vs he or she needs. To obtain weekly fruit and vegetable servings consumption, the number of times per week F&Vs are consumed will be multiplied by the number of servings consumed each time. Serving size will be age adjusted. To assess sugar sweetened beverage (SSB) consumption, mothers will be asked questions from an adapted version of the Pre-School-Aged Beverage Intake Questionnaire (BEVQ-15) in addition to items developed by the study team and based on previous studies conducted by the co-investigators.
Group differences in children's physical activity levels as assessed by accelerometry. | 18 months-24 months postpartum
  Child's PA will be measured objectively using accelerometry. We will use the Actical accelerometer (formerly MiniMitter Co, Philips Respironics, Bend, OR), a small waterproof device (28x27x10mm) weighing 17g, which is omnidirectional (sensing motion in all planes), and integrates the degree and intensity of motion. We will use procedures co-investigators have used successfully in previous studies of young adolescents, toddlers and their mothers, placing the accelerometer on the non-dominant ankle with a non-removable, reinforced hospital band worn next to the skin, under socks, for 7 consecutive days. Accelerometers will be attached on the day of the 18- and 24-month assessment battery and removed one week later. Data will be collected in 1-minute epochs. The time-stamped data will be examined. Summary statistics will include average and total activity counts and minutes in moderate to vigorous physical activity (MVPA)
Group differences in children's reported physical activity, screen time and other sedentary activities over time as assessed by the Child Physical Activity Assessment. | 2 weeks-24 months postpartum
  This 14-item self-report assessment includes questions about tummy time, crawling, walking, sedentary behavior and screen time for infants and toddlers. Questions were compiled based on a body of literature related to assessing infant/toddler physical activity.
Group differences in children's mean BMI z-scores over time as assessed through child weight and length measurements over time. | 2 weeks-24 months postpartum
  Child weight (to the nearest ounce) and recumbent length (to the nearest 1/8 inch) will be measured using a digital scale and a recumbent measuring board (in accordance with IHS guidelines). All measurements will be taken in triplicate, removing the most disparate measurement, and averaging the remaining two. Averages will be used to calculate BMI z-scores using age- and sex-specific World Health Organization (WHO) Child Growth Standards.

SECONDARY OUTCOMES:
Group differences in levels of maternal stress over time as assessed by the Perceived Stress Scale 4 (PSS-4). | <32 weeks gestation-24 months postpartum
  Completed by mothers, the 4-item questionnaire will assess maternal stress. This 4-item scale is scored with a 5-point Likert scale. The range of the 5-point Likert scale is as follows: 0 (never), 1 (almost never), 2 (sometimes), 3 (fairly often), 4 (very often). We will reverse scores for items 2 and 3. On these questions, the scores will be as follows: 4 (never), 3 (almost never), 2 (sometimes), 1 (fairly often), 0 (very often). Scores for each item will be summed to get a total score. The lowest score is 0 and the highest score is 16. Higher scores are correlated to more stress (worse outcome).
Group differences in depression scores over time as assessed by the Centers for Epidemiological Studies Depression Scale-Revised-10 (CESDR-10). | <32 weeks gestation-24 months postpartum
  The 10-item questionnaire is a validated adapted version of the CESD-R (which has been utilized to assess depression with Navajo mothers) to screen for depression in adolescents. The questionnaire asks participants to rate how often over the past two weeks have they experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling sad. Response options range from 0 to 4 for each item, with 0 = not at all or less than 1 day in the last 2 weeks, 1 = 1-2 Days, 2 = 3-4 Days, 3 = 5-7 Days, 4 = Nearly every day for 2 weeks. Scores for each item will be summed to get a total score. Scores range from 0 to 40, with high scores indicating greater depressive symptoms (worse outcome). A CESD-R score of 8 or greater indicates individuals at risk for clinical depression.
Group differences in alcohol and drug use over time as assessed by the Alcohol, Smoking and Substance Involvement Screening Test (ASSIST). | <32 weeks gestation-24 months postpartum
  Adapted from WHO ASSIST questionnaire covering 10 main substance groups, this 15-item questionnaire screens for all levels of problem or risky substance use (alcohol, illegal drugs, and prescription drugs). A risk score is provided for each substance, and scores are grouped into low, moderate, or high risk. Only items 2-7 and 9-14 are scored. Each question has a set of responses to choose from and each response has a numerical score. The scores from questions 2-7 and questions 9-14 are added together to produce an ASSIST risk score for each substance that falls into 1 of 3 categories: low, moderate, or high substance-related risk. Participants with risk scores 3 or less are at lower risk of problems related to their substance use. Participants scoring between 4 and 26 are at moderate risk and may be experiencing some of these problems right now. A score of 27 or higher for any substance suggests that the participant is at high risk of dependence/dependent on that substance.
Group differences in how infant biologic measures of metabolic health at delivery and 6 months postpartum correlate to maternal biologic measures of metabolic health. | Delivery-6 months postpartum
  Blood specimens will be collected from mothers at delivery and 6 months postpartum. Blood specimens will be collected from infants at delivery (cord blood), 6 and 12 months postpartum. Laboratory testing will be completed to assess levels of fasting glucose, insulin, HOMA-IR, leptin, adiponectin, lipids panels, and c-reactive protein in mothers and babies to examine how infant metabolic health relates to maternal metabolic health at delivery, and whether there are between group differences in this relationship over time. In all cases, higher levels indicate poorer metabolic health.
Group differences in infant metabolic health at delivery, 6 and 12 months postpartum. | Delivery-12 months postpartum
  Blood specimens will be collected from infants at delivery (cord blood), 6 and 12 months postpartum. Laboratory testing will be completed to assess levels of fasting glucose, insulin, HOMA-IR, leptin, adiponectin, lipids panels, and c-reactive protein in infants to examine whether there are between group differences in infant metabolic health at delivery and over time (delivery to 12 months postpartum). In all cases, higher levels indicate poorer metabolic health. In addition, results will be used to determine whether infants are insulin resistant and/or leptin insensitive (these will be dichotomous outcomes) and between group differences will be assessed at delivery and over time (delivery to 12 months postpartum).
Examination of whether group differences in infant metabolic health at delivery, 6, 12 months postpartum are moderated/mediated by sociodemographic, biological (pre-pregnancy BMI, etc), and psychosocial characteristics of mothers at baseline. | Delivery-12 months postpartum
  Blood specimens will be collected from infants at delivery (cord blood), 6 and 12 months postpartum. Laboratory testing will be completed to assess levels of fasting glucose, insulin, HOMA-IR, leptin, adiponectin, lipids panels, and c-reactive protein in infants. In all cases, higher levels indicate poorer metabolic health. Analyses will be conducted to determine whether between group differences in metabolic health at delivery and over time (delivery to 12 months postpartum) are moderated or mediated by sociodemographic, biological, and psychosocial characteristics of mothers at baseline.
Examination of how the COVID-19 pandemic impacted infant/child feeding practices, food and water security, and study participation. | 32 weeks gestation - 24 months postpartum
  All primary outcomes will be examined pre- and post- COVID-19 to determine how the COVID-19 pandemic impacted these outcomes with and without intervention. Describe food-related and non food-related stressors mothers experienced due to the COVID-19 pandemic. Examine how these stressors impacted breastfeeding and mothers' feeding and parenting practices. Examine how study participation and curriculum dosage changed during the COVID-19 pandemic. Examine demographic differences/similarities between participants who could be reached by remote intervention/control lessons and assessments vs. those who could not be reached. Study outcomes will provide important knowledge about how future home-visiting interventions can best adapt to community-level crises.
Explore how and why the COVID-19 pandemic impacted infant/child feeding practices, food and water security, and study participation (with a subset of 25% of participants). | 12 months postpartum - 36 months postpartum
  Qualitative interviews will be conducted with 25% of study participants. Sample will be stratified water security, study group, and site. Describe how and why the COVID-19 pandemic impacted infant/child feeding practices, food and water security, and study participation through extraction of primary themes from in-depth interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Barlow, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (3):
- United States (3):
  - Johns Hopkins Center for American Indian Health, Fort Defiance, Arizona
  - Johns Hopkins Center for American Indian Health, Whiteriver, Arizona
  - Johns Hopkins Center for American Indian Health, Shiprock, New Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ingalls A, Rosenstock S, Foy Cuddy R, Neault N, Yessilth S, Goklish N, Nelson L, Reid R, Barlow A. Family Spirit Nurture (FSN) - a randomized controlled trial to prevent early childhood obesity in American Indian populations: trial rationale and study protocol. BMC Obes. 2019 May 6;6:18. doi: 10.1186/s40608-019-0233-9. eCollection 2019. PMID 31080627